CLINICAL TRIAL: NCT04421131
Title: mHealth-supported Telecolposcopy for Cervical Cancer Programs in Low-resource Settings: Evaluation (mIVAA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Pro00100618; R21TW011223-02 (NIH)
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Results first posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-09

CONDITIONS: Cervical Cancer
Keywords: cervical cancer screening; colposcopy; digital health
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- mIVAA (Experimental): Screened for cervical cancer with mIVAA in mobile units
  Interventions: Device: Pocket colposcope/Mobile phone camera; Other: mIVAA

INTERVENTIONS:
Device: Pocket colposcope/Mobile phone camera — The Pocket colposcope or mobile phone camera will be used to capture magnified digital images of the cervix
Other: mIVAA — A mobile-phone-based telemedicine platform that enables remote consultation with an expert colposcopist

SUMMARY:
The central hypothesis is that use of mIVAA (mobile Inspección Visual con Ácido Acético - Spanish for Visual Inspection with Acetic Acid (VIA)) will increase the proportion of VIA positive women who complete follow-up clinical evaluation compared to VIA positive women in situations in which mIVAA was not used, thus potentially improving cervical cancer treatment and survival rates. The study will collect qualitative and quantitative data to examine the feasibility and preliminary impact of mIVAA on reducing attrition for follow-up clinical evaluations.

DETAILED DESCRIPTION:
The study will be conducted in Lima, Peru in the context of mobile units operated by La Liga for promoting cancer screening. mIVAA comprises two components: a digital imaging device and a telemedicine platform.

1. The digital imaging device is either a mobile phone camera or the pocket colposcope plugged into a mobile phone.
2. The telemedicine platform is mobile phone-based, with an interface for midwives in the mobile units to enter patient information and acquire and upload cervical images, and an interface for the colposcopists based remotely to review the cervical images and patient information and return feedback.

The specific aim is to pilot test mIVAA in a community-based setting in Peru.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Patients coming to the mobile unit for cervical cancer screening
* Willing to allow use of mIVAA during screening with VIA.
* Agree to be audio recorded

Exclusion Criteria:

* Currently pregnant
* History of hysterectomy
* Does not understand the study purpose and details
* Is not willing to sign an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lavanya Vasudevan, PhD, Principal Investigator — Duke University
Locations (1):
- La Liga Contra el Cancer-Peru, Lima, Peru

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Informed consent was obtained prior to establishing eligibility. One consented participant was deemed ineligible and one was ineligible due to not completing screening.
Groups:
- mIVAA (Mobile Inspección Visual Con Ácido Acético - Spanish for Visual Inspection With Acetic Acid): Screened for cervical cancer with mIVAA in mobile units
  Pocket colposcope/Mobile phone camera: The Pocket colposcope or mobile phone camera will be used to capture magnified digital images of the cervix
  mIVAA: A mobile-phone-based telemedicine platform that enables remote consultation with an expert colposcopist
Period: Overall Study
Arm/Group | mIVAA (Mobile Inspección Visual Con Ácido Acético - Spanish for Visual Inspection With Acetic Acid)
Started | 110
Referred to a Follow up Screening | 17
Completed | 102
Not Completed | 8
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 2
Not completed — App crashed | 5

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Arm/Group | mIVAA (Mobile Inspección Visual Con Ácido Acético - Spanish for Visual Inspection With Acetic Acid)
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 102
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 3
  More than one race | 78
  Unknown or Not Reported | 16
Region of Enrollment [Count of Participants; unit: Participants]
  Peru | 102

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Women Referred to a Follow up Screening Appointment With a Colposcopist Who Did Not Attend the Appointment
Time Frame: up to 142 days
Population: Participants who were referred.
Measure: Number; unit: percentage of women
Arm/Group | mIVAA (Mobile Inspección Visual Con Ácido Acético - Spanish for Visual Inspection With Acetic Acid)
Number analyzed (Participants) | 17
percentage of women | 82.4

2. Secondary Outcome: Percentage of Women Approached Who Consented to Participate in Study
Time Frame: up to 142 days
Population: Women who were approached to participate in the study.
Measure: Number; unit: percentage of women
Arm/Group | mIVAA (Mobile Inspección Visual Con Ácido Acético - Spanish for Visual Inspection With Acetic Acid)
Number analyzed (Participants) | 112
percentage of women | 100

3. Secondary Outcome: Percentage of Women Approached Who Refused to Participate in Study
Time Frame: up to 142 days
Population: Women who were approached to participate in the study.
Measure: Number; unit: percentage of women
Arm/Group | mIVAA (Mobile Inspección Visual Con Ácido Acético - Spanish for Visual Inspection With Acetic Acid)
Number analyzed (Participants) | 112
percentage of women | 0

4. Secondary Outcome: Number of Visual Inspection With Acetic Acid (VIA) Screened Women Who Are VIA+
Description: Women who screened positive (i.e., suspicious) for cervical cancer/pre-cancer.
Time Frame: up to 142 days
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | mIVAA (Mobile Inspección Visual Con Ácido Acético - Spanish for Visual Inspection With Acetic Acid)
Number analyzed (Participants) | 102
Participants | 6

5. Secondary Outcome: Average Number of Days From Screening to When a Follow up Appointment is Scheduled
Time Frame: up to 142 days
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | mIVAA (Mobile Inspección Visual Con Ácido Acético - Spanish for Visual Inspection With Acetic Acid)
Number analyzed (Participants) | 102
days | 26.6 (41.1)

6. Secondary Outcome: Median Number of Days From Screening to When a Follow up Appointment is Scheduled
Time Frame: up to 142 days
Population: Participants who completed the study.
Measure: Median (Full Range); unit: days
Arm/Group | mIVAA (Mobile Inspección Visual Con Ácido Acético - Spanish for Visual Inspection With Acetic Acid)
Number analyzed (Participants) | 102
days | 6 [3 to 116]

7. Secondary Outcome: Percentage of Women Who Were Screened Using mIVAA
Time Frame: up to 142 days
Measure: Number; unit: percentage of women
Arm/Group | mIVAA (Mobile Inspección Visual Con Ácido Acético - Spanish for Visual Inspection With Acetic Acid)
Number analyzed (Participants) | 102
percentage of women | 100

8. Secondary Outcome: Average Number of Hours From Screening to When Expert Enters Feedback Using mIVAA
Time Frame: up to 142 days
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | mIVAA (Mobile Inspección Visual Con Ácido Acético - Spanish for Visual Inspection With Acetic Acid)
Number analyzed (Participants) | 102
hours | 2.0 (5.89)

9. Secondary Outcome: Percentage of mIVAA Screened Women With Expert Feedback Within 0-7 Days of mIVAA Screening Date
Time Frame: up to 7 days
Population: Participants who completed the study.
Measure: Number; unit: percentage of women
Arm/Group | mIVAA (Mobile Inspección Visual Con Ácido Acético - Spanish for Visual Inspection With Acetic Acid)
Number analyzed (Participants) | 102
percentage of women | 100

10. Secondary Outcome: Number of Women Screened Positive (i.e., Suspicious) for Cervical Cancer/Pre-cancer by Midwife
Time Frame: up to 142 days
Measure: Count of Participants; unit: Participants
Arm/Group | mIVAA (Mobile Inspección Visual Con Ácido Acético - Spanish for Visual Inspection With Acetic Acid)
Number analyzed (Participants) | 102
Participants | 6

11. Secondary Outcome: Number of Women Screened Positive (i.e., Suspicious) for Cervical Cancer/Pre-cancer by Expert Colposcopist
Time Frame: up to 142 days
Measure: Count of Participants; unit: Participants
Arm/Group | mIVAA (Mobile Inspección Visual Con Ácido Acético - Spanish for Visual Inspection With Acetic Acid)
Number analyzed (Participants) | 102
Participants | 17

12. Secondary Outcome: Average Number of Attempts Per Woman Before a Readable Image is Obtained by Midwife
Time Frame: up to 142 days
Measure: Mean (Standard Deviation); unit: attempts
Arm/Group | mIVAA (Mobile Inspección Visual Con Ácido Acético - Spanish for Visual Inspection With Acetic Acid)
Number analyzed (Participants) | 102
attempts | 3.35 (0.7)

13. Secondary Outcome: Percentage of mIVAA Screened Women With at Least 1 Image Rated as Readable by Expert
Time Frame: up to 142 days
Measure: Number; unit: percentage of women
Arm/Group | mIVAA (Mobile Inspección Visual Con Ácido Acético - Spanish for Visual Inspection With Acetic Acid)
Number analyzed (Participants) | 102
percentage of women | 84.3

14. Secondary Outcome: Number of Instances of Network Failure
Time Frame: up to 142 days
Measure: Number; unit: network failures
Arm/Group | mIVAA (Mobile Inspección Visual Con Ácido Acético - Spanish for Visual Inspection With Acetic Acid)
Number analyzed (Participants) | 102
network failures | 1

ADVERSE EVENTS:
Time Frame: Up to 142 days
Arm/Group | mIVAA (Mobile Inspección Visual Con Ácido Acético - Spanish for Visual Inspection With Acetic Acid)
All-Cause Mortality (participants affected / at risk) | 0/110
Serious Adverse Events (participants affected / at risk) | 0/110
Other Adverse Events (participants affected / at risk) | 0/110

LIMITATIONS AND CAVEATS:
In March of 2021, NIH agreed to reduce the scope of the study. Therefore, the investigators did not conduct any Aim 2 study activities indicated in the Study Protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT04421131/Prot_SAP_000.pdf